CLINICAL TRIAL: NCT02205632
Title: Relationships Between Macular Pigment Optical Density and Lacquer Cracks in High Myopic Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None
Other Study IDs: MPSII-RMB
Record Dates: First submitted 2014-07-22; First posted 2014-07-31 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: High Myopia

ARMS (2):
- High myopic patients with lacker craks (Other)
  Interventions: Device: MPS II
- High myopic patients without lacker cracks (Other)
  Interventions: Device: MPS II

INTERVENTIONS:
Device: MPS II

SUMMARY:
Lutein ans zeaxanthin, carotenoids provided by dietary intake are mainly located in the macular area.

Its absorption peak at 460 nm may reduce photic damages. The macular pigment density can be evaluated by its optical density.

Reduced macular pigment level is a significant risk factor for age-macular degeneration. The nutritional intake can minimise the risk of age-macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years-old
* High axial myopia < -6 dioptries
* Presence or not of lacquer cracks in Bruch's membrane in one or both eyes
* Patients with social security coverage

Exclusion Criteria:

* Age <18 years-old
* Amblyopia in the studied eye
* Prior ocular surgery
* Corneal disease or severe dry eye syndrome
* Other retinal disease: diabetic retinopathy, age-related macular degeneration, macular hole, epiretinal membrane central
* Extensive chorioretinal atrophy
* Allergy to tropicamide
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Association between lacquer cracks related to high myopia and the macular pigment optical density | 1 day

SECONDARY OUTCOMES:
The macular pigment optical density among high myopic patients | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas LEVEZIEL, MD, PhD, Principal Investigator — Poitiers University Hospital
Locations (1):
- ophthalmology department, Poitiers University Hospital, Poitiers, Vienne, France